CLINICAL TRIAL: NCT01368224
Title: PLACEBO-CONTROLLED STUDY OF THE EFFECT OF TWO FOOD SUPPLEMENTS ON SKIN REACTIVITY
Brief Title: Two Supplemented Against Skin Reactivity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: L'Oreal (Industry)
Collaborators: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Audrey Gueniche, L'Oreal
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1040341
Record Dates: First submitted 2011-06-06; First posted 2011-06-07 (Estimated); Last update posted 2011-06-07 (Estimated); Status verified 2011-06

CONDITIONS: Skin Sensitivity; Trans-epidermal Water Loss; Clinical Score; Assessment of Skin Moisturization Factors; Assessment of Serum Immune-regulatory Cytokine; Evaluation of Intestinal Flora Composition
Keywords: Skin sensitivity; Trans-epidermal water loss; Clinical score; skin moisturization factors; serum immune-regulatory cytokine; Evaluation of intestinal flora composition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Maltodextrin (Placebo Comparator)
  Interventions: Dietary Supplement: Lactobacillus paracasei NCC 2461 and Bifidobacterium longum NCC3001
- Lactobacillus paracasei NCC 2461 (ST 11) (Experimental): 1x1010 CFU of Lactobacillus paracasei NCC 2461 (ST 11)
  Interventions: Dietary Supplement: Lactobacillus paracasei NCC 2461 and Bifidobacterium longum NCC3001
- Lactobacillus paracasei+ Bifidobacterium longum (Experimental): 1x1010 CFU of Lactobacillus paracasei NCC 2461 (ST 11) + 1x1010 CFU of Bifidobacterium longum (NCC3001)
  Interventions: Dietary Supplement: Lactobacillus paracasei NCC 2461 and Bifidobacterium longum NCC3001

INTERVENTIONS:
Dietary Supplement: Lactobacillus paracasei NCC 2461 and Bifidobacterium longum NCC3001 — 1 treatment unit, in the form of a sachet of powder, to be reconstituted in a glass of water and taken once daily for 8 weeks (from D1 to D57), except if the last visit is bring forward or put back for no more than 3 days, in which case the subject will continue treatment until the final visit.
  Oral route.

SUMMARY:
In recent decades, the incidence of subjects presenting reactive skin has considerably increased in industrialized countries. Probiotics are live microorganisms which, when ingested in sufficient amounts, have beneficial effects on human health. The mechanism underlying the effect of probiotics involves, in part, regulation of the composition and/or metabolic activity of the intestinal microbiota.. It is postulated that following interaction of probiotics with the intestinal epithelium, associated intestinal cells become activated and consequently mediators are released into the blood circulation. Mediators, activated intestinal epithelial cells and possibly bacterial fractions might reach the skin through the bloodstream where they potentially could exert effects.The objective of this study was to assess the effects of probiotics on reactive skin symptoms. The strain Lactobacillus paracasei NCC2461 was tested alone and in combination with the strain Bifidobacterium longum NCC3001 in a randomized, double-blind study. The two strains were selected for their immune-modulatory properties demonstrated in in vitro and other preclinical studies as well as in a pilot clinical trial.

Ninety-six women presenting reactive skin were randomized to 3 groups: placebo (n = 32), L. paracasei NCC2461 alone (n = 32) and L. paracasei NCC2461 + B. longum NCC3001 (n = 32). The supplements were administered by the oral route for 58 days (1010 CFU/day).

The objective of the clinical trial was to determine, in vivo, the effect of food supplements on reactive skin symptoms (as measured by skin sensitivity and the reconstruction of barrier function post-repeated tape stripping).

The secondary objectives were to determine the effect of the food supplements on leg skin dryness and facial skin roughness and the associated biochemical, immunological and microbiological factors.

Accordingly, the subjects' skin sensitivity was determined by the capsaicin test. The reconstruction of barrier function was determined by measuring the trans-epidermal water loss (TEWL) post-repeated stripping using a SERVOMED evaporimeter. A clinical score for skin dryness and roughness was assigned by a dermatologist. The subjects also assessed their leg and facial skin dryness themselves. Each analysis was conducted at the various time points.

In parallel, assessment of the skin moisturizing factors and serum inflammatory and immune-regulatory cytokines were performed. Finally, key components of the intestinal microbiota were analyzed.

DETAILED DESCRIPTION:
The probiotics and particularly Lactobacillus paracasei and Bifidobacterium longum are of value with respect to the homeostasis of dry and sensitive skin.

An initial study (study report No. 1020813, DERMSCAN dated 2/10/2004) showed that the combination of L. paracasei NCC2461 (ST11) with Bifidobacterium lactis NCC2818 (Bb12) induced an improvement in certain parameters related to skin reactivity. However, the probiotics have not been tested separately.

It was thus considered important to conduct a clinical trial aiming at confirming and documenting the data generated by the previous study and, also determining the specific efficacy of L. paracasei NCC2461 (ST11) on reactive skin symptoms. The latter probiotic strain was selected on the basis of its proven immune-modulatory properties (scientific dossier ST11-Nestec Benyacoub and Gueniche. Scientific evidence supporting the use of Lactobacillus paracasei NCC2461 (ST11) for Innéov. Report 11.02.2005 and references 23, 24, 31-33). The strain was combined or not with a probiotic of the Bifidobacterium genus, particularly Bifidobacterium longum NCC3001. The data generated by various preclinical studies (NRC in-house studies) and clinical studies (public) show that this probiotic strain is able to modulate immune mechanisms and could interfere with inflammatory reactions.

Moreover, the probiotic combination concept enables providing potential benefit all along the gastrointestinal tract, inducing maintenance of an optimum intestinal flora.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject.
* Gender: female.
* Subject aged more than 18 years and less than 35 years (inclusive)
* Phototype: I to IV
* Caucasian race.
* For women of child-bearing potential, effective contraception for at least 12 weeks and maintained throughout the study and for 1 month after completion of the study.
* Sensitive skin: (1) as per the subjective evaluation questionnaire in appendix 12.2. (with at least 1 positive response to one of the first 3 questions) and (2) responder to the capsaicin test at one of the 3 lowest concentrationsSubject known to have dry leg skin (clinical score of at least 2 as per the scale).
* Subject known to have rough cheek skin (clinical score of at least 3 as per the scale).
* Low consumers of fermented dairy products (less than 125 g/d) and agreeing not to eat fermented dairy products containing live bacteria (yogurt, cottage cheese, fermented dairy products, unpasteurized cheese, etc.) for the duration of the study.

Exclusion Criteria:

* Post-menopausal woman.
* Pregnant or breast-feeding woman or woman planning pregnancy during the study.

  --Volunteer with a skin disease in the test areas (particularly acne rosacea). Volunteer presenting a stable or progressive serious disease (investigator's assessment).
* Immunocompromised subject.
* Subject allergic to one of the constituents of the test products and, in particular, capsaicin or pepper.
* Alcohol intake greater than 2 glasses of wine daily or 1 glass of liquor daily.
* Smoker of more than 6 cigarettes/day.
* Subject presenting excessive exposure to sunlight or UV radiation (investigator's assessment).
* Subjects regularly practicing aquatic or nautical sports.
* Subjects regularly attending a sauna.
* Subject with cardiovascular or circulatory history.
* Subject with a history of skin cancer or malignant melanoma.
* Subject with a history of intestinal surgery.
* Intake of antibiotics, corticosteroids, non-steroidal anti-inflammatories or immune-suppressants.
* Subject practicing sports for more than 5 hours per week.
* Subject having taken mineral or vitamin supplements in the 3 months preceding the study (investigator's assessment).
* Lacto-ovo-vegetarian, vegetarian.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2004-06; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
skin sensitivity and skin barrier reconstruction
  determining the effect of food supplements on skin reactivity (measured by skin sensitivity and the skin barrier function reconstruction after repeated tape-stripping).

SECONDARY OUTCOMES:
dryness , roughness, biochemical factors and safety
  * determining the effect of the food supplements on leg skin dryness and facial skin roughness,
  * determining the effect of the food supplements on the associated biochemical and immunological factors,
  * Evaluating the safety of the study products.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric BOUDJEMA, MD, Principal Investigator — Dermscan
Locations (1):
- DERMSCAN - PharmaScan, Villeurbanne, France